CLINICAL TRIAL: NCT01468779
Title: Effect of the Probiotics Use in Patients Undergoing Surgery for Periampullary Neoplasia - A Randomized Clinical Trial
Brief Title: Effect of Probiotics in Patients Undergoing Surgery for Periampullary Neoplasms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: FIPE - Fundo de Incentivo a Pesquisa do Hospital de Clínicas de Porto Alegre (Unknown); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Heloisa Sommacal, nutritionist, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 09256; HCPA09256 (Other: 09-256)
Record Dates: First submitted 2011-08-03; First posted 2011-11-09 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Periampullary Carcinoma Nos
Keywords: Periampullary cancer; Surgery; Dietary supplementation; Nutritional assessment
MeSH Terms: interventions — Probiotics; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): The patients submitted to periampullary cancer surgery will receive sugar pills in the preoperative and postoperative period.
  Interventions: Dietary Supplement: Sugar pill
- Probiotics (Active Comparator): The probiotics pills are given orally in the amount of two pills twice a day as early as two days before surgery until ten days after surgery.
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — The probiotics pills are given orally in the amount of two pills twice a day as early as two days before surgery until ten days after surgery.
  Arms: Probiotics
Dietary Supplement: Sugar pill
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to evaluate the effect of the probiotic use in patients with periampullary cancers undergone curative or palliative treatment considering nutritional status, postoperative complications, infection rate, length of hospitalization and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of surgery for periampullary cancer

Exclusion Criteria:

* Patients submitted to periampullary surgery without pathologic confirmation of cancer
* Patients unwilling to be a part of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Mortality | participants will be followed for the duration of hospital stay, an expected average of 15 days
  Death will be considered as the primary outcome related to complications of surgical treatment in postoperative period

SECONDARY OUTCOMES:
Postoperative infection rate | participants will be followed for the duration of hospital stay, an expected average of 15 days
  To assess postoperative infection rate in patients submitted to periampullary cancer surgery using probiotics.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- See also: Related Info — http://www.hcpa.ufrgs.br/content/view/1596/1117/